CLINICAL TRIAL: NCT06486012
Title: Regular Use of Antibacterial Photodynamic Therapy in the Management and Prevention of Periodontitis Symptoms in Diabetic Patients - Special Attention to Diabetic Balance and Metabolism
Brief Title: Regular Use of aPDT in the Management and Prevention of Periodontitis Symptoms in Diabetic Patients
Acronym: APDT-T2D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wellbeing Services County of Pirkanmaa (Other)
Collaborators: Tampere University (Other); University of Helsinki (Other); Mehiläinen Health Care Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R24021L
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2; Pre-diabetes; Periodontal Diseases; Periodontitis
Keywords: periodontitis; diabetes; T2D; aPDT; aMMP-8
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Periodontal Diseases; Periodontitis; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Randomized clinical study on a medical device.
Who Masked: Outcomes Assessor
Masking Description: Data will be collected using individual study codes for participants. Study codes do not reveal which group the participant has belonged to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Standard oral hygiene and home-use of Lumoral Treatment aPDT device.
  Interventions: Device: Lumoral Treatment; Other: Standard oral hygiene
- Control group (Active Comparator): Standard oral hygiene
  Interventions: Other: Standard oral hygiene

INTERVENTIONS:
Device: Lumoral Treatment — Photodynamic antibacterial dual-light device home-use with a marker substance
  Arms: Study group
Other: Standard oral hygiene — Standard oral hygiene performed at home

SUMMARY:
This is an investigator-initiated clinical study to establish easy referral and access for diabetic patients from primary health care to oral health care facilities for preventive oral care, periodontal assessment, and treatment, and to investigate the impact of regular home use of aPDT medical device on plaque control and gingival health, when used as an adjunct treatment to standard oral hygiene, and the effect on diabetes control in patients with the risk of periodontal disease, compared to a standard home care oral hygiene regimen.

DETAILED DESCRIPTION:
In earlier studies, a bi-directional link between diabetes and periodontitis has been established: high glucose levels increase the risk of periodontitis while glycemic control is likely to worsen with untreated periodontitis. The treatment of diabetic patients should include easy access from diabetes clinics to oral health care facilities to reduce the potential risks of periodontal disease, or deterioration of existing symptoms of periodontal disease. As part of a holistic approach to healthcare and its resources, more attention needs to be paid to the early detection, and prevention of oral diseases in diabetic patients. Novel testing and treatment methods can play a key role, and a good collaboration between diabetes and oral health care facilities is essential.

The aMMP-8 test can be used to assess the risk of periodontal disease. If the test is positive, latent MMP-8 is activated, so the inflammatory cascade is activated and provides real-time information. The test can also be used to monitor the success of the treatment outcome and can be used to determine the interval between maintenance treatments. In addition, patients' oral self-care should be improved, as most of the work in preventing oral diseases is done at home. The home use of photodynamic dual light therapy (aPDT) can provide additional benefits and also engage patients not only in self-care but also in the whole treatment process. Preliminary studies show that aPDT improves the treatment and maintenance outcomes, and potentially reduces the risk of periodontal disease in addition to self-care.

The combination of easy access to treatment could have wide benefits individually, and also at the community level, including the possibility of building a cost-effective preventive care pathway for patients with prediabetes, type 2 diabetes, and periodontitis, and identifying the risks of both diseases and treating already detected diseases early and in a timely manner.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patient treated at community health care;
* At least 18 years old;
* Presence of ≥20 teeth;
* Agreement to participate in the study, and to sign a written consent form;
* Ability to cooperate with the treatment protocol according to coordinator investigator's assessment.

Exclusion Criteria:

* Oral thrush;
* Known sensitivity to near-infrared or antibacterial blue light.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Bleeding on probing (BOP) | 12 months
  Change in bleeding on probing (BOP) A full-mouth assessment at six sites per tooth (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) Gingival bleeding is considered as positive if bleeding occurs within 15 seconds after gentle probing with a probe at the sulcus Dichotomous scoring to each site of the tooth as bleeding "1 present" and "0 absent" BOP is reported as the percentage (%) of sites with positive findings Calculation formula: number of bleeding sites/ 6 times number of teeth

SECONDARY OUTCOMES:
Visual Plaque Index (VPI) | 6 months
  Assessment of six index teeth, measured at four sites per tooth:
  * Dichotomous scoring to each site of the tooth as plaque "1 present" and "0 absent"
  * VPI reported as the percentage (%) of sites with plaque
  * Calculation formula: number of sites with plaque/ 4 times number of teeth
Visual Plaque Index (VPI) | 12 months
  Assessment of six index teeth, measured at four sites per tooth:
  * Dichotomous scoring to each site of the tooth as plaque "1 present" and "0 absent"
  * VPI reported as the percentage (%) of sites with plaque
  * Calculation formula: number of sites with plaque/ 4 times number of teeth
Periodontal Pocket Depth (PPD) | 6 months
  A full-mouth assessment, measured at six sites per tooth. Assessed from the base of the pocket to the gingival margin (mm)
Periodontal Pocket Depth (PPD) | 12 months
  A full-mouth assessment, measured at six sites per tooth. Assessed from the base of the pocket to the gingival margin (mm)
Clinical Attachment Level (CAL) | 6 months
  A full-mouth assessment, measured at six sites per tooth
  Assessed as the distance from the cementoenamel junction (CEJ) to the bottom of the periodontal pocket (mm)
  To calculate CAL, two measurements are needed: distance from the gingival margin to the CEJ and PPD; in recession: PPD + gingival margin to the CEJ; in tissue overgrowth: PPD - gingival margin to the CEJ
Clinical Attachment Level (CAL) | 12 months
  A full-mouth assessment, measured at six sites per tooth
  Assessed as the distance from the cementoenamel junction (CEJ) to the bottom of the periodontal pocket (mm)
  To calculate CAL, two measurements are needed: distance from the gingival margin to the CEJ and PPD; in recession: PPD + gingival margin to the CEJ; in tissue overgrowth: PPD - gingival margin to the CEJ
Active matrix metalloproteinase 8 (aMMP-8) | 6 months
  The oral rinse fluid sample collection and the aMMP-8 marker analysis will be performed using Periosafe test (Dentognostics GmbH) according to the manufacturer's instructions.
Active matrix metalloproteinase 8 (aMMP-8) | 12 months
  The oral rinse fluid sample collection and the aMMP-8 marker analysis will be performed using Periosafe test (Dentognostics GmbH) according to the manufacturer's instructions.
Periodontopathic bacteria | 6 months
  Quantification of periodontopathic bacteria by 16S rRNA sequencing analysis.
  Microbiological samples can be collected using Iso Taper Paper Points, size-20 (VDW GmbH) from selected gingival/periodontal pockets with maximum initial probing depth. The paper points can be placed into sterile, small-aliquot containers, and immediately stored at -20°C until analysis
Periodontopathic bacteria | 12 months
  Quantification of periodontopathic bacteria by 16S rRNA sequencing analysis.
  Microbiological samples can be collected using Iso Taper Paper Points, size-20 (VDW GmbH) from selected gingival/periodontal pockets with maximum initial probing depth. The paper points can be placed into sterile, small-aliquot containers, and immediately stored at -20°C until analysis
Metabolomics | 12 months
  Nuclear magnetic resonance (NMR) -based metabolomics analysis for biomarkers that include 39 clinically validated routine markers to explore connections between metabolites and an individual's health status.
hsCRP | 12 months
  Diagnosis and monitoring of latent inflammation. High-sensitivity CRP tests can determine slight changes to CRP levels within the CRP normal range, which would otherwise be missed by standard tests. Hs-CRP tests can help identify more specific issues and chronic inflammation over the long term.
LPS | 12 months
  Gram-negative bacteria-derived lipopolysaccharides (LPS) are known to be associated with various negative health effects. Activity of serum lipopolysaccharides will be measured with Limulus Amebocyte Lysate assay from 1:5 diluted serum samples at 405 nm as an end-point assay

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Heikkinen, Professor, Principal Investigator — Wellbeing Services of County Pirkanmaa
Locations (1):
- Wellbeing Services of County Pirkanmaa, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmad R, Haque M. Oral Health Messiers: Diabetes Mellitus Relevance. Diabetes Metab Syndr Obes. 2021 Jul 1;14:3001-3015. doi: 10.2147/DMSO.S318972. eCollection 2021. PMID 34234496
- [Background] Choi SE, Sima C, Pandya A. Impact of Treating Oral Disease on Preventing Vascular Diseases: A Model-Based Cost-effectiveness Analysis of Periodontal Treatment Among Patients With Type 2 Diabetes. Diabetes Care. 2020 Mar;43(3):563-571. doi: 10.2337/dc19-1201. Epub 2019 Dec 27. PMID 31882408
- [Background] Gasner NS, Schure RS. Periodontal Disease. 2025 May 12. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554590/ PMID 32119477
- [Background] Kononen E, Gursoy M, Gursoy UK. Periodontitis: A Multifaceted Disease of Tooth-Supporting Tissues. J Clin Med. 2019 Jul 31;8(8):1135. doi: 10.3390/jcm8081135. PMID 31370168
- [Background] Nazir MA. Prevalence of periodontal disease, its association with systemic diseases and prevention. Int J Health Sci (Qassim). 2017 Apr-Jun;11(2):72-80. PMID 28539867
- [Background] Liccardo D, Cannavo A, Spagnuolo G, Ferrara N, Cittadini A, Rengo C, Rengo G. Periodontal Disease: A Risk Factor for Diabetes and Cardiovascular Disease. Int J Mol Sci. 2019 Mar 20;20(6):1414. doi: 10.3390/ijms20061414. PMID 30897827
- [Background] Pakarinen S, Saarela RKT, Valimaa H, Heikkinen AM, Kankuri E, Noponen M, Alapulli H, Tervahartiala T, Raisanen IT, Sorsa T, Patila T. Home-Applied Dual-Light Photodynamic Therapy in the Treatment of Stable Chronic Periodontitis (HOPE-CP)-Three-Month Interim Results. Dent J (Basel). 2022 Nov 2;10(11):206. doi: 10.3390/dj10110206. PMID 36354651
- [Background] Salminen A, Maatta AM, Mantyla P, Leskela J, Pietiainen M, Buhlin K, Suominen AL, Paju S, Sattler W, Sinisalo J, Pussinen PJ. Systemic Metabolic Signatures of Oral Diseases. J Dent Res. 2024 Jan;103(1):13-21. doi: 10.1177/00220345231203562. Epub 2023 Nov 15. PMID 37968796
- See also: Bashir, N.Z., Singh, HA. & Virdee, S.S. Indocyanine green-mediated antimicrobial photodynamic therapy as an adjunct to periodontal therapy: a systematic review and meta-analysis. Clin Oral Invest 25, 5699-5710 (2021). — https://doi.org/10.1007/s00784-021-03871-2
- See also: Berger, V., Bour, L., Carter, K. et al. A roadmap to using randomization in clinical trials. BMC Med Res Methodol 21, 168 (2021). — https://doi.org/10.1186/s12874-021-01303-z
- See also: Borgnakke, W.S., Poudel, P. Front. Dent. Med, Volume 2 - 2021. Diabetes and Oral Health: Summary of Current Scientific Evidence for Why Transdisciplinary Collaboration Is Needed. — https://doi.org/10.3389/fdmed.2021.709831
- See also: Centers for Disease Control and Prevention (CDC), July 2023. Periodontal Disease. — https://www.cdc.gov/oral-health/about/gum-periodontal-disease.html
- See also: Sorsa, T, Nwhator, SO, Sakellari, D, Grigoriadis, A, Umeizudike, KA, Brandt, E, Keskin, M, Tervahartiala, T, Pärnänen, P, Gupta, S, Mohindra, R, Bostanci, N, Buduneli, N, Räisänen, IT. Front. Oral Health, 10 June 2022, Sec. Oral Infections and Microbes — https://doi.org/10.3389/froh.2022.897115
- See also: World Health Organization (WHO). Diabetes, Oct 2023. Newsroom, Fact sheets, Detail, Diabetes. — https://www.who.int/news-room/fact-sheets/detail/diabetes
- See also: Zhang Y., Leveille S.G., Shi L., Camhi S.M. Disparities in Preventive Oral Health Care and Periodontal Health Among Adults With Diabetes. Prev Chronic Dis 2021;18:200594 — http://dx.doi.org/10.5888/pcd18.200594